CLINICAL TRIAL: NCT01426074
Title: A Phase II/Pharmacodynamic Study of Preoperative or Definitive FOLFOX Plus Bevacizumab, With the Additional Pharmacodynamic Goal of Assessing Tumor Blood Flow as Measured by Dynamic Contrast-enhanced MRI, and the Induction of Hypoxia and Apoptosis as Measured by PET in Patients With Rectal Cancer
Brief Title: DCE-MRI PET Bevacizumab Study in Rectal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: UPCC 05209
Record Dates: First submitted 2011-08-29; First posted 2011-08-31 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Rectal Cancer Patients
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Bevacizumab 5 mg/kg — Intravenously every two weeks

SUMMARY:
This study will determine the following: the response rate (including pathological CR rate), TTP, and complications of treatment in patients with rectal cancer treated with FOLFOX bevacizumab, the alteration of tumor blood flow (assessed by DCE-MRI as percentage change in Ktrans) after 1 cycle of bevacizumab therapy compared to baseline value in patients treated with FOLFOX alone and those treated with bevacizumab at 5 mg/kg., the degree of hypoxis (measured by tumor uptake of the 2-nitroimidazole EF5) induced by bevacizumab treatment and its relationship to changes in tumor blood flow, and the degree of apoptosis (measured by tumor uptake of di-annexin V) induced by bevacizumab treatment and its relationship to changes in tumor blood flow.

DETAILED DESCRIPTION:
The primary objectives of this study will determine the following: the response rate (including pathological CR rate), TTP, and complications of treatment in patients with rectal cancer treated with FOLFOX bevacizumab, the alteration of tumor blood flow (assessed by DCE-MRI as percentage change in Ktrans) after 1 cycle of bevacizumab therapy compared to baseline value in patients treated with FOLFOX alone and those treated with bevacizumab at 5 mg/kg., the degree of hypoxis (measured by tumor uptake of the 2-nitroimidazole EF5) induced by bevacizumab treatment and its relationship to changes in tumor blood flow, and the degree of apoptosis (measured by tumor uptake of di-annexin V) induced by bevacizumab treatment and its relationship to changes in tumor blood flow. The secondary objectives of this study is to determine in an exploratory fashion the relationship between tumor blood flow, hypoxia induction, and apoptosis induction , and time to progression in patients continuing on to receive Bevacizumab 5 mg/kg, to analyze archival tumor from the patients treated in this trial for mutations in the MKK7 and SEK1 genes, and by semi-quantitative IHC for these and other relevant proteins, to determine the relationship between vascular proliferation as measured by DCE-MRI and markers of endothelial cell proliferation, and to obtain pilot data on whether assays that measure vascular endothelial cell mitogenic stimulation and mitogenic activity may predict response to therapy, time to progression and overall survival in patients receiving bevacizumab 5 mg/kg.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically documented advanced or metastatic adenocarcinoma of the rectum, T3 or T4, N any, M0 or M1. Patients must have available and identified tissue for immunohistochemical analysis and agree to submit it for the correlative endpoints. When available, formalin-fixed,paraffin-embedded tissue from previous biopsy or surgical resection will suffice.
* Patients must measurable disease as defined by the RECIST criteria as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20mm with conventional techniques on either CT, MRI, or EUS. marker (CEA) elevation alone is in sufficient for entry.
* Patients may have had prior adjuvant treatment of rectal cancer. The prior treatment regimen must not have included bevacizumab but may have included oxaliplatin and the last dose of chemotherapy must have been > 6 months prior to study entry. Patients with prior radiotherapy are acceptable. It must be at least 2 weeks since administration of radiation therapy and all signs of toxicity must have abated.
* Patients with prior malignancies other than colorectal cancer are allowed, provided they have been treated with curative, intent, and have no evidence of recurrence of that malignancy.
* Patients must be age 18 years or older.
* Patients must have an ECOG performance status of 0-1.
* The following required required Initial Laboratory Values should be obtained within 4 weeks of the start of treatment:

Granulocytes ≥ 1,500/ml Platelet Count ≥ 100,000/ml Creatinine ≤ 1.5 x upper limit of normal Bilirubin ≤ 1.5 x upper limit of normal AST ≤ 5 x upper limit of normal Urine: Urine protein: creatinine ration ≤ 1.0 at screening

* Patients must not be pregnant or lactating as chemotherapy is though to present substantial risk to the fetus/infant
* Patients must have a life expectancy of greater than three months.
* Patients must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients may not be receiving any other investigational agents.
* Patients with the following contraindication to MRI are excluded: Hypersensitivity to gadolinium Contraindicated metallic device, including pacemaker, non-MRI compatible aneurysm clip, other non-MRI compatible mechanical and/or electrical device, or metallic fragments.
* Patients with severe claustrophobia
* Patients with a history of allergic reactions attributed to Flagyl (metronidazole) which has a chemical structure similar to EF5 are excluded.
* Patients with T1 or T2 N0M0 disease are not eligible.
* Major surgical procedure, open biopsy or significant traumatic injury within 28 days to Day 0, anticipation of need for major surgical procedure during the course of the study. Minor surgical procedures such as port placement, fine needle aspirations or core biopsies within 3 days prior to Day 0.
* Patients with serious nonhealing wounds, ulcers, or bone fractures.
* Patients with a history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 0.
* Patients with a history of myocardial infarction, unstable angina, or cerebrovascular accident < 6 months prior to registration.
* Patients with clinically significant peripheral vascular disease.
* Patients with New York Heart Association Class II or greater congestive heart failure (Class II is defined as symptoms of fatigue, dyspnea or other symptoms with ordinary physical activity) See Appendix E.
* Patients using oral or parenteral anticoagulation are not excluded provided they are on a stable dose of anticoagulant.
* patients with pre-existing hypertension should be on a stable antihypertensive regimen and have a blood pressure ≤ 150/100 mmHg at the time of enrollment.
* Patients must not have known brain metastases because the study drug has not been adequately tested in this setting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2014-06-11 (Actual); Study Completion 2014-06-11 (Actual)

PRIMARY OUTCOMES:
Pathologic Complete Response (pCR)

CONTACTS AND LOCATIONS:
Overall Officials: Peter O'Dwyer, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine